CLINICAL TRIAL: NCT05464940
Title: Impact of Intravenous Caffeine on Atrial Electrical Properties and Potential Arrythmia Induction in Patients With Paroxysmal Atrial Fibrillation: The COFFEE-AF Trial
Brief Title: Impact of Intravenous Caffeine on Atrial Electrical Properties and Potential Arrythmia Induction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute, Overland Park, KS (Unknown); Texas Cardiac Arrhythmia Institute, Austin, TX, USA (Unknown); Loma Linda University, Loma Linda, California, USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KCHRRF-COFFEE AF-0012
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The COFFEE-AF (How caffeine Induces Atrial Tachyarrhythmias) trial will be a multi-center, randomized, double-blinded trial of intravenous caffeine versus placebo among patients undergoing pulmonary vein isolation procedures for AF.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group assigned to receive caffeine (Active Comparator)
  Interventions: Other: Intravenous caffeine
- Group assigned to receive masked placebo (Placebo Comparator)
  Interventions: Other: Masked Placebo

INTERVENTIONS:
Other: Intravenous caffeine — Group assigned to receive caffeine will receive intravenous(IV) caffeine and sodium benzoate infusion starting at 250-500 mg.
  This method will use an automated algorithm that adjusts the flow of the infusion depending on the individual's sex and weight and then in a serial fashion in response to blood caffeine measurements. Serial blood caffeine measurements at pre-determined intervals according to the algorithm will be until a steady state is obtained.
  Arms: Group assigned to receive caffeine
Other: Masked Placebo — The patients assigned to the masked placebo will receive 5% dextrose in 0.45% saline using the same infusion protocol for a random length of time that was within 1 standard deviation(SD) of the mean time to achieve a steady state using the caffeine protocol (17+4 min).
  To maintain blinding, caffeine blood concentration measurements that will be randomly generated within 2 SDs of the predicted values calculated by the algorithm will be used and verbally communicated for placebo infusions.
  Arms: Group assigned to receive masked placebo

SUMMARY:
This "How caffeine Induces Atrial Tachyarrhythmias" trial will be a multi-center, randomized, double-blinded trial of intravenous caffeine versus placebo among patients undergoing pulmonary vein isolation procedures for Atrial Fibrillation(AF).

DETAILED DESCRIPTION:
The mechanism by which caffeine might change cardiac electrophysiologic properties is largely unknown. Most of the prior studies conducted have evaluated the correlation based on the premise of oral consumption. One caveat among such study designs can be underreporting or overreporting the amount of caffeine ingested. To this date, no clinical trials exist that has studied the in vivo effects of caffeine to assess the atrial refractory period and conduction velocity and its potential to cause atrial or ventricular ectopy or sustained arrythmia induction including Atrial Tachycardia(AT)/Atrial Fibrillation(AF)/Ventricular Tachycardia(VT)/Ventricular Fibrillation(VF). As it is hypothesized that decreasing the atrial refractory period can render atria more prone to fibrillation. The pulmonary veins have proven integral to AF pathophysiology, the relationship between pulmonary vein electrophysiology and lifestyle factors in particular has not previously been assessed. It is also not clear if caffeine increases the risk of AF on those patients with known AF diagnosis. To bridge this gap, a randomized controlled trial is proposed to assess the effects of intravenous caffeine on atrial activity during AF ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

All adult patients from 21-90 years of age with new onset Paroxysmal Atrial Fibrillation presenting in sinus rhythm or AF of recent onset (the latter confirmed by sinus rhythm documented no more than 1 week prior) undergoing AF ablation will be included in the study.

Exclusion Criteria:

Patients will be excluded if any of the following were identified:

1. History of substance abuse or alcoholism.
2. Left ventricular ejection fraction <50%.
3. Liver dysfunction.
4. Pregnancy.
5. Inability to give informed consent.
6. Amiodarone uses within 1 month prior to procedure.
7. AAD use within 24 h prior to the procedure
8. Severe intolerance to caffeine.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Atrial Fibrillation Induction | 1 day
  Induction of Atrial fibrillation will be attempted by pacing and isoproterenol infusion following study drug infusion. The ability to induce atrial fibrillation (yes or no) will be recorded as the primary outcome.

SECONDARY OUTCOMES:
Number of patients with Site-specific changes in AERP(Atrial Effective Refractory Period) | 1 day
  It helps assess changes in AERP in milli-seconds at different potential trigger points of Atrial fibrillation during the procedure.
Number of patients with Changes in conduction time | 1 day
  Changes in conduction time is the changes in conduction of electrical impulses with caffeine during the procedure.
Number of patients with Induction of Atrial Fibrillation/Atrial Tachycardia (AF/AT) or other arrhythmias | 1 day
  By infusing caffeine, intraprocedural for stimulation and detection of potential triggers of ablation, will caffeine infusion lead to the start of atrial fibrillation (AF), atrial tachycardia(AT) or any other arrhythmias.
Number of patients with Identification of non-pulmonary triggers of AF | 1 day
  Identification of non-pulmonary triggers of AF

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (9):
- United States (9):
  - Loma Linda University, Loma Linda, California
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center Clinic, Independence, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Texas Cardiac Arrythmia Institute, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCarthy DM, Mycyk MB, DesLauriers CA. Hospitalization for caffeine abuse is associated with abuse of other pharmaceutical products. Am J Emerg Med. 2008 Sep;26(7):799-802. doi: 10.1016/j.ajem.2007.10.018. PMID 18774047
- [Background] Chen Y, Parrish TB. Caffeine's effects on cerebrovascular reactivity and coupling between cerebral blood flow and oxygen metabolism. Neuroimage. 2009 Feb 1;44(3):647-52. doi: 10.1016/j.neuroimage.2008.09.057. Epub 2008 Oct 19. PMID 19000770
- [Background] Temple JL. Caffeine use in children: what we know, what we have left to learn, and why we should worry. Neurosci Biobehav Rev. 2009 Jun;33(6):793-806. doi: 10.1016/j.neubiorev.2009.01.001. Epub 2009 Jan 20. PMID 19428492
- [Background] Reissig CJ, Strain EC, Griffiths RR. Caffeinated energy drinks--a growing problem. Drug Alcohol Depend. 2009 Jan 1;99(1-3):1-10. doi: 10.1016/j.drugalcdep.2008.08.001. Epub 2008 Sep 21. PMID 18809264
- [Background] Wendt IR, Stephenson DG. Effects of caffeine on Ca-activated force production in skinned cardiac and skeletal muscle fibres of the rat. Pflugers Arch. 1983 Aug;398(3):210-6. doi: 10.1007/BF00657153. PMID 6634380
- [Background] Rashid A, Hines M, Scherlag BJ, Yamanashi WS, Lovallo W. The effects of caffeine on the inducibility of atrial fibrillation. J Electrocardiol. 2006 Oct;39(4):421-5. doi: 10.1016/j.jelectrocard.2005.12.007. Epub 2006 Aug 21. PMID 16919674
- [Background] Bodar V, Chen J, Gaziano JM, Albert C, Djousse L. Coffee Consumption and Risk of Atrial Fibrillation in the Physicians' Health Study. J Am Heart Assoc. 2019 Aug 6;8(15):e011346. doi: 10.1161/JAHA.118.011346. Epub 2019 Aug 5. PMID 31378120
- [Background] Larsson SC, Drca N, Jensen-Urstad M, Wolk A. Coffee consumption is not associated with increased risk of atrial fibrillation: results from two prospective cohorts and a meta-analysis. BMC Med. 2015 Sep 23;13:207. doi: 10.1186/s12916-015-0447-8. PMID 26394673
- [Background] Conen D, Chiuve SE, Everett BM, Zhang SM, Buring JE, Albert CM. Caffeine consumption and incident atrial fibrillation in women. Am J Clin Nutr. 2010 Sep;92(3):509-14. doi: 10.3945/ajcn.2010.29627. Epub 2010 Jun 23. PMID 20573799